CLINICAL TRIAL: NCT00154596
Title: Etiology Study of Kawasaki Disease--A Prospective Household and Case Control Study
Brief Title: Etiology Study of Kawasaki Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 930004318
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Kawasaki Disease
Keywords: etiology; transmission; vasculitis; household; etiology of disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Vasculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, throat swab, nasopharyngeal aspiration, and rectal swab will be obtained during acute illness and at convalescence (about 2 weeks after discharge). These specimens will be processed for viral isolation, bacterial culture and toxin detection, PCR, subtractive cloning, VIDISCA, gene chips, peptide library, cytokine/chemokine measurement, antibody detection for specific pathogens, etc. Questionnaire for contact history and clinical symptoms will be performed.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the infectious etiology of Kawasaki disease (KD); a prospective household and case control study for Kawasaki disease will be done. The investigators will enroll Kawasaki disease cases who have at least five of the following manifestations:

1. fever for over 5 days
2. neck lymphadenopathy
3. lip fissure and/or strawberry tongue
4. skin rash
5. nonpurulent bulbar conjunctivitis
6. palm/sole erythema and induration followed by desquamation, or coronary artery aneurysm with less than 5 of the above manifestations (atypical Kawasaki disease)

The KD cases will receive virological (virus isolation from the blood, throat swabs and rectal swabs or stool, gene chip for possible viruses from stored RNA and DNA), bacterial (blood, throat swabs and stool: bacterial culture and stored strain for further toxin or superantigen detection), and serological (Mycoplasma pneumoniae, Chlamydiae pneumoniae, ASLO, HHV6, EV71, peptide library approach for auto-antibody or pathogen-related antibody, stored serum for further workup) workup. Stored DNA from the blood will also be performed.

DETAILED DESCRIPTION:
Patient Selection and Family Surveillance: At National Taiwan University Hospital in Taiwan, we will study patients who fulfill the criteria of Kawasaki disease or atypical Kawasaki disease and their household family members from 2004 to Dec 2005. Institutional Review Board approval will be obtained for this study and informed consents will be obtained from all subjects or their parents. If patients at the emergent service, outpatient clinic or inpatient ward had clinical syndromes suggestive of EV71 infection, they and their household family members were asked to participate in the study. Throat and rectal swabs for virus isolation, and the first blood sample. Clinical manifestations, courses and outcomes were recorded. If at any point the patients suspected of infection displayed clinical symptoms, the other family members in the same household were asked to undergo screening by virus isolation of throat swabs, and received the first blood sample. Questionnaire-based interviews were used to collect information including demographic data, the number of bedrooms in the household, contact time, pattern and presence of current/recent signs and symptoms (cough, rhinorrhea, sore throat, rash, fever, abdominal pain and diarrhea) and preceding contact history with extra-household people who had clinical illness. Follow-up telephone interviews repeated questions about signs and symptoms at 2, 4 and 8-week intervals. If any household family member reported experiencing signs or symptoms suggestive of Kawasaki disease during the follow-up period, the household member will receive further clinical assessment and repeated laboratory investigation for Kawasaki disease. A second blood sample was obtained from the KD cases and all their household family members 4 weeks after the first blood sample was obtained. Control case selection: An age- and sex-matched control will be randomly selected. The control will be the admitted patients in the same ward who have other diagnoses (such as pneumonia, UTI, tonsillitis). They will also receive the screen for virus and bacterial workup as the household members do.

Definitions of Kawasaki disease and atypical Kawasaki disease:

1. Criteria for Kawasaki disease:

   * equal to or over five of the following: fever for more than 5 days, non-purulent conjunctivitis, skin rash, palm/sole induration and erythema followed by desquamation, neck lymphadenopathy, strawberry tongue or lip fissure/bleeding
2. Atypical Kawasaki disease; less than five of the above but with coronary artery aneurysm.

Laboratory Methods

1. Virus Isolation and Serotyping:

   Throat swabs, rectal swabs or stool samples were submitted for virus isolation. Samples were inoculated into human embryonic fibroblast, LLC-MK2, HEp-2 and rhabdomyosarcoma (RD) cell cultures. When cytopathic effect involved more than 50% of the cell monolayer, cells were scraped and subjected to indirect fluorescent antibody staining with specific antibodies (Chemicon International Inc., Temecula, CA) or typed by specific methods according to the suspected types of viruses.
2. Molecular diagnosis for viruses or other pathogens difficult to be cultivated:

   1. Viral RNA and RNA extraction: RNA and DNA extraction will be performed by using Isolation Kit according to the manufacturer's guide. (RNA extraction kit, Qiagen). 140 uL of throat swab was mixed with AVL buffer for 10 to 15 minutes at room temperature. Then, spin down the mixture. Add 560 uL 100% alcohol into the pellet and incubated for at least 10 minutes at room temperature. The mixture will be put into the spin column and centrifuged at 8000 rpm for 1 minute twice. Then, 500uL of AW1 buffer will be added and the mixture will be centrifuged at 80000 rpm for 1 minute, and then 500uL of AW2 buffer will be added and centrifuged at 14000 rpm for 3 minutes. Discard the solution and centrifuge at 14000 rpm for 2 minutes. Finally, 25 to 30 uL of AVE buffer will be added and centrifuged at 8000 to 10000 rpm for 1 minute.
   2. Reverse transcription: RT will be performed with 1st strand cDNA Synthesis Kit for RT-PCR (Roche). Mix the previously extracted RNA with reagents including buffer, MgCl2, dNTP, Oligo-p(dT)15 primer, RNase inhibitor, reverse transcriptase, briefly vortex, incubate the reaction at 25oC for 10 minutes and then 42oC for 60 minutes. Finally incubate at 99oC for 5 minutes and then cool to 4oC for 5 minutes.
   3. Real-time TagMan PCR for enterovirus, adenovirus or other viral etiology. The primers and probes for enterovirus and other virus real time PCR are in the following table. Primers and probes for PanEV were selected based on highly conserved regions in the 5'-untranslated region of the enterovirus genome. The primers and probes for EV71 were selected based on the most diverse and specific genetic regions in the VP1 region of the enterovirus genome. Other potential viruses, such as adenovirus, or other respiratory viruses will also be performed by PCR or RT-PCR or real-time PCR following the rules of the above procedures.
   4. Representational differential analysis followed by subtractive cloning
3. Bacterial cultures and toxin detection: Cultures were obtained from the pharynx, and rectum of patients with acute KD before the start of the immune globulin intravenous infusion and from control patients with the use of a Baxter Diagnostics Culturette system that contains a cotton swab. The primary data collection sheet was completed and held at the site where specimens were obtained. The plates were then examined for all â-hemolytic group A streptococci and all S aureus that were coagulase positive by the tube test. These isolates were then screened in a blinded fashion for the presence of bacterial superantigen production by immunodiffusion with antisera against known staphylococcal and streptococcal superantigens as described previously. (Lee PK and Schlieveret PM).
4. Serological test: Serological tests for antibody detection of Mycoplasma pneumoniae, Chlamydiae pneumoniae, ASLO will be measured by commercial kits. Neutralizing antibody for enterovirus will be performed by standard protocol of the neutralization test on microtiter plates. EV71 isolate TW/2272/98 was amplified and purified as an antigen for m-capture ELISA for EV71 IgM Detection. If potential pathogen is defined, further serology test for the specific pathogen will be done later.
5. Statistical Analysis: Data were analyzed with the SAS Statistical Package (Version 8.2, SAS Institute, Cary, North Carolina). We used Student's t test for continuous variables and c 2 test for categorical data. After univariate analysis screened statistically significant variables, forward stepwise multiple logistic regression analysis was performed to adjust confounders simultaneously and to calculate multivariate-adjusted odds ratios. The level of model selection was set at 0.15 for in-and-out models. P < .05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill the criteria of Kawasaki disease or atypical Kawasaki disease and their household family members

Exclusion Criteria:

* Not cases of Kawasaki disease

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We will enroll Kawasaki disease cases who have at least five of the following manifestations: 1) fever for over 5 days, 2) neck lymphadenopathy, 3) lip fissure and/or strawberry tongue, 4) skin rah, 5) nonpurulent bulbar conjunctivitis, 6) palm/sole erythema and induration followed by desquamation, or cases with coronary artery aneurysm but less than 5 of the above manifestations (atypical Kawasaki disease).
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2004-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Viral infections associated with Kawasaki disease | 2014/3
  The mean age of the 226 KD cases was 2.07 years, and the male to female ratio was 1.43 (133 boys to 93 girls). Their mean fever duration was 7.5 days with a mean peak temperature of 39.7°C. In addition to the typical symptoms of fever, neck lymphadenopathy, lip fissure and/or strawberry tongue, skin rash, nonpurulent bulbar conjunctivitis, palm/sole erythema, and induration followed by periungual desquamation, these KD cases also exhibited cough (69%), rhinorrhea (58%), and diarrhea (45%). Cases of KD had a significantly higher positive rate of viral isolation in comparison with the control group (7.5% vs. 2.2%, p = 0.02). Compared with the control group, cases of KD were more likely to have overall positive rates of viral PCR (50.4% vs. 16.4%, p < 0.001) and for various viruses including enterovirus (16.8% vs. 4.4%, p < 0.001), adenovirus (8.0% vs. 1.8%, p = 0.007), human rhinovirus (26.5% vs. 9.7%, p < 0.001), and coronavirus (7.1% vs. 0.9%, p = 0.003).

CONTACTS AND LOCATIONS:
Overall Officials: Luan-Yin Chang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Result] Chang LY, Chiang BL, Kao CL, Wu MH, Chen PJ, Berkhout B, Yang HC, Huang LM; Kawasaki Disease Research Group. Lack of association between infection with a novel human coronavirus (HCoV), HCoV-NH, and Kawasaki disease in Taiwan. J Infect Dis. 2006 Jan 15;193(2):283-6. doi: 10.1086/498875. Epub 2005 Dec 2. PMID 16362893
- [Result] Chang LY, Lu CY, Shao PL, Lee PI, Lin MT, Fan TY, Cheng AL, Lee WL, Hu JJ, Yeh SJ, Chang CC, Chiang BL, Wu MH, Huang LM. Viral infections associated with Kawasaki disease. J Formos Med Assoc. 2014 Mar;113(3):148-54. doi: 10.1016/j.jfma.2013.12.008. Epub 2014 Feb 1. PMID 24495555
- [Result] Tsai HC, Chang LY, Lu CY, Shao PL, Fan TY, Cheng AL, Hu JJ, Yeh SJ, Chang CC, Huang LM. Transmission of acute infectious illness among cases of Kawasaki disease and their household members. J Formos Med Assoc. 2015 Jan;114(1):72-6. doi: 10.1016/j.jfma.2014.07.005. Epub 2014 Sep 6. PMID 25205598
- [Result] Lee YC, Kuo HC, Chang JS, Chang LY, Huang LM, Chen MR, Liang CD, Chi H, Huang FY, Lee ML, Huang YC, Hwang B, Chiu NC, Hwang KP, Lee PC, Chang LC, Liu YM, Chen YJ, Chen CH; Taiwan Pediatric ID Alliance; Chen YT, Tsai FJ, Wu JY. Two new susceptibility loci for Kawasaki disease identified through genome-wide association analysis. Nat Genet. 2012 Mar 25;44(5):522-5. doi: 10.1038/ng.2227. PMID 22446961